CLINICAL TRIAL: NCT00001284
Title: Structural and Functional Imaging of Neuropsychiatric Patients and Normal Volunteers With 1.5 Tesla MRI
Brief Title: Magnetic Resonance Imaging (MRI) of Neuropsychiatric Patients and Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 910124; 91-M-0124
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-02-25

CONDITIONS: Genotype; Allelic Frequencies of Genetic Markers; Brain Mapping; Brain Disease; fMRI
Keywords: Cognition; Schizophrenia; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Dopaminergic Mechanisms
MeSH Terms: conditions — Brain Diseases; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to use brain imaging technology to compare differences in brain structure, chemistry, and functioning in individuals with brain and mental disorders compared to healthy volunteers.

Schizophrenia is a brain disorder that results from subtle changes and abnormalities in neurons. These deficits likely occur in localized regions of the brain and may result in widespread, devastating consequences. The neuronal abnormalities are inherited through a complex combination of genetic and environmental factors. Brain imaging technologies can be used to better characterize brain changes in individuals with schizophrenia. This study will use magnetic resonance imaging (MRI) scans to identify predictable, quantifiable abnormalities in neurophysiology, neurochemistry and neuroanatomy that characterize schizophrenia and other neurological and neuropsychiatric disorders....

DETAILED DESCRIPTION:
This protocol is meant to provide a matrix for multiple, simultaneous brain imaging investigations using magnetic resonance imaging (MRI). We intend to study regional brain structure, physiology, and biochemistry in living human subjects, both healthy and ill. Based on multiple clinical, neuropathological, and functional neuroimaging studies, it is clear that schizophrenia is a brain disorder arising from subtle neuronal deficits (for lack of more specific terminology). These deficits likely arise in a few key regions such as dorsolateral prefrontal cortex and hippocampal formation, that result in widespread, multifaceted, and devastating clinical consequences. These neuronal deficits are clearly heritable, although in a complex fashion from multiple genes interacting in an epistatic fashion with each other and the environment. We hypothesize that these neuronal deficits, clearly resulting in quantifiable behavioral abnormalities in schizophrenic patients, will produce predictable, quantifiable aberrations in neurophysiology that we can "map" using magnetic resonance imaging. In spite of numerous functional imaging findings, clinical applications remain scarce and pathognomic findings absent. Therefore, we do not anticipate that an approach based solely on any one modality is likely to significantly advance our knowledge base. Instead, we propose to create brain imaging datasets for individual human subjects predicated on 1) the appraisal of brain function from multiple domains simultaneously; 2) the characterization of brain function via summation and intercorrelation of these data; and 3) the digestion of these data based on the parsing of complex clinical phenomenology into quantifiable neurophysiological parameters. Thus, in addition to the identification of those parameters that best characterize and identify manifest schizophrenia (i.e., state variables), we hypothesize that some of these fundamental characteristics will be heritable. These fundamental characteristics, so-called endo- or intermediate phenotypes, represent powerful tools to find susceptibility genes and have already generated a number of linkage findings.

ELIGIBILITY:
* INCLUSION CRITERIA:

CONTROLS:

No psychiatric or severe chronic medical illness at the time of the study, and by history. This includes the absence of substance abuse histories, learning disabilities and all DSM IV disorders. The investigators will evaluate medical histories and medical conditions that are judged not to interfere with the study may be allowed.

No use of psychotropic substances in the last 3 months.

There is no upper age limit. The lower age limit is 18 years.

PATIENTS:

Schizophrenia, any subtype or schizoaffective disorder according to DSM IV, as detailed in protocol # 89-M-0160 ("Inpatient Evaluation of Neuropsychiatric Inpatients") and #95-M-0150 ("A Longitudinal Investigation of Siblings of Schizophrenic and Manic-Depressive Patients").

Bipolar Disorder with Psychotic Features according to DSM IV as detailed in protocol.

Menstrually-Related Mood Disorder.

Mild to Moderate Parkinson's Disease (Hoehn and Yahr Stage 1-3).

EXCLUSION CRITERIA:

CONTROLS AND PATIENTS:

Impaired hearing.

Pregnancy.

Head trauma with loss of consciousness in the last year, or any evidence of functional impairment due to and persisting after head trauma.

Patients or healthy volunteers with a known risk from exposure to high magnetic fields (e.g. patients with pace makers) and those who have metallic implants (e.g. braces) in the head region (likely to create artifact on the MRI scans) will be excluded from participating in the fMRI studies.

Patients:

Coexistence of another major mental illness at the time of the study. If the patients experienced other mental illnesses in the past (e.g. major depression), then this should be judged to be fully recovered.

Criteria for substance abuse met in the last 6 months.

Criteria for substance dependence in the last year. If criteria for dependence were met in the past, then the duration of the disorder was less than 3 years, or not judged to have produced long-term brain changes to allow the patient to be in the study.

Major concurrent medical illness likely to interfere with the acquisition of the task.

Concomitant medications which could interfere with performance on the task.

Presence of dyskinetic movements of the face and tongue (likely to interfere with eyeblink measures, or of gross involuntary movements of the whole body (likely to interfere with positioning in the MRI scanner).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2802 (Actual)
Dates: Start 1991-05-10; Study Completion 2019-02-25

PRIMARY OUTCOMES:
Brain Activation | Per MRI Scan

CONTACTS AND LOCATIONS:
Overall Officials: Karen F Berman, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Belliveau JW, Kennedy DN Jr, McKinstry RC, Buchbinder BR, Weisskoff RM, Cohen MS, Vevea JM, Brady TJ, Rosen BR. Functional mapping of the human visual cortex by magnetic resonance imaging. Science. 1991 Nov 1;254(5032):716-9. doi: 10.1126/science.1948051.
- [Background] Ogawa S, Tank DW, Menon R, Ellermann JM, Kim SG, Merkle H, Ugurbil K. Intrinsic signal changes accompanying sensory stimulation: functional brain mapping with magnetic resonance imaging. Proc Natl Acad Sci U S A. 1992 Jul 1;89(13):5951-5. doi: 10.1073/pnas.89.13.5951. PMID 1631079
- [Background] Kwong KK, Belliveau JW, Chesler DA, Goldberg IE, Weisskoff RM, Poncelet BP, Kennedy DN, Hoppel BE, Cohen MS, Turner R, et al. Dynamic magnetic resonance imaging of human brain activity during primary sensory stimulation. Proc Natl Acad Sci U S A. 1992 Jun 15;89(12):5675-9. doi: 10.1073/pnas.89.12.5675. PMID 1608978